CLINICAL TRIAL: NCT05314322
Title: The Impacts of Deep Brain Stimulation on Dual-task Gait Performance in Parkinson's Disease: Focusing on Long-term Outcome and the Effects of Stimulation Modes
Brief Title: Deep Brain Stimulation on Dual-task Gait Performance in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-02-016A
Record Dates: First submitted 2022-03-16; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Dual-task walking; Executive function
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency group (Experimental): Deep brain stimulation's parameter: Frequency adjusted to 130Hz, with other parameters fixed
  Interventions: Procedure: Deep brain stimulation with high frequency
- Low frequency group (Experimental): Deep brain stimulation's parameter: Frequency adjusted to 60Hz, with other parameters fixed
  Interventions: Procedure: Deep brain stimulation with low frequency

INTERVENTIONS:
Procedure: Deep brain stimulation with high frequency — Deep brain stimulation implanted at the patients' Substantia Nigra
  Arms: High frequency group
Procedure: Deep brain stimulation with low frequency — Deep brain stimulation implanted at the patients' Substantia Nigra
  Arms: Low frequency group

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease after Alzheimer's disease. Motor symptoms include rigidity, bradykinesia, tremor, and postural instability, these motor symptoms can cause gait dysfunction. Non-motor symptoms include depression, dysarthria, cognitive disability, and sleep disturbance. Although these symptoms can be improved through drug treatment, when the course of PD reaches the middle to late stage, it will still face the situation of weakened drug efficacy and the drug side effects increased. When medication can no longer adequately control the motor symptoms of PD, deep brain stimulation (DBS) becomes a powerful option. DBS is a surgical treatment that involves implanting one or more electrodes into specific areas of the brain, which deliver electrical stimulation to regulate or destroy abnormal neural signal patterns in the target area. The effect of DBS has been proven whether it is in improving motor-related symptoms or non-motor-related symptoms, but there are still some areas that have not been compared before and after the surgery, such as: gait variability, executive functions and dual-task walking. In addition, the parameters of electrical stimulation for DBS will also affect the clinical characteristics of patients. Due to the large difference between individual cases, the recommendation of the electrical stimulation frequency still not be established. Therefore, the influence of DBS and its parameters on the symptoms of PD is a topic worthy of discussion. Purposes: (1) To investigate the long-term effects of DBS on the symptoms of PD. (2) To investigate the effects of DBS stimulation frequencies on walking performance and executive function in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Age: 50~80 yrs old
* Hoehn and Yahr stage ≤ IV after DBS operation
* Implanted DBS system for at least 6 months
* MMSE ≥24

Exclusion Criteria:

* Other neurological disorders
* Any major systemic, psychiatric, visual, and musculoskeletal disturbances or other causes of walking inability

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task gait performance: Stride length | Three days after frequency adjustment
  Using the OPTO gait system to evaluate stride length
Dual-task gait performance: Double limb support time | Three days after frequency adjustment
  Using the OPTO gait system to evaluate double limb support time
Executive function - Inhibition control | Three days after frequency adjustment
  Using the Stroop test to evaluate inhibition control
Executive function - Shifting attention | Three days after frequency adjustment
  Using the Trail Making Test to evaluate shifting attention
Executive function - Working memory | Three days after frequency adjustment
  Using the Digit span test to evaluate working memory
Cognitive function | Every 6-month up to 2 years
  Using the Montreal Cognitive Assessment (MoCA) to evaluate cognitive function
Non-motor symptoms | Every 6-month up to 2 years
  Using the Non-motor Symptoms Scale (NMSS) to non-motor symptoms

SECONDARY OUTCOMES:
Usual gait performance: Stride length | Three days after frequency adjustment
  Using the OPTO gait system to evaluate stride length
Usual gait performance: Double limb support time | Three days after frequency adjustment
  Using the OPTO gait system to evaluate double limb support time
Brain activity: Prefrontal Cortex | Three days after frequency adjustment
  Using Functional near-infrared spectroscopy (fNIRS) to evaluate brain activity of Prefrontal Cortex with the formula: Hb diff=HbO-HbR
Brain activity: Supplementary Motor Cortex | Three days after frequency adjustment
  Using Functional near-infrared spectroscopy (fNIRS) to evaluate brain activity of Supplementary Motor Area with the formula: Hb diff=HbO-HbR
Brain activity: Premotor Cortex | Three days after frequency adjustment
  Using Functional near-infrared spectroscopy (fNIRS) to evaluate brain activity of Premotor Cortex with the formula: Hb diff=HbO-HbR
Functional activity: Gait and balance performance | Every 6-month up to 2 years
  Using the Timed up and go test to evaluate functional activity
Functional activity: Lower limb function | Every 6-month up to 2 years
  Using the 30s Chair Stand Test to evaluate functional activity
Balance performance | Every 6-month up to 2 years
  Using the Mini-BEST test to evaluate balance performance
Motor symptoms | Every 6-month up to 2 years
  Using the Unified Parkinson's Disease Rating Scale (UPDRS) part 3 to evaluate motor symptoms
Parkinson's Disease patients' Quality of life | Every 6-month up to 2 years
  Using the Parkinson's Disease Questionnaire (PDQ-39) evaluate quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided